CLINICAL TRIAL: NCT01739153
Title: Effect of Cheese on Cardiovascular Risk
Acronym: ECCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); Dairy Research Institute (Other); Dairy Farmers of Canada (Other); Centre National Interprofessionel de l'Economie Laitière (Other); Dairy Australia (Industry); Nederlandse Zuivel Organisatie (Other)
Responsible Party: Principal Investigator, Arne Astrup, Prof., MD, Head of Department, Department of Nutrition, Exercise and Sports, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B302
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Hyperlipidemia
Keywords: Dairy; Cheese; Blood lipid concentrations; Blood lipid sizes; Fecal fat; Fat digestibility; bile acids
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CARB diet (Experimental): The CARB diet will be a low-fat diet where cheese is replaced by starchy carbohydrates and lean meat. The CARB diet will have the same protein content (15 E%) and quality as the CHEESE and MEAT diet but a lower fat content (approx. 25 E%) and a correspondingly higher carbohydrate content (approx. 60 E%).
  Interventions: Other: Dietary intervention: CARB (High Carbohydrate intake)
- CHEESE diet (Experimental): The CHEESE diet will contain cheese in amounts corresponding to 120 g/day on a 10 MJ diet (approx. 1.8 MJ from cheese). A high dose of cheese is chosen to provoke effects within this short time frame. The cheese types used in this study will be Danbo (45+) and Cheddar (50+) which will be supplied in equal amounts. The CHEESE diet will have the same macronutrient composition as that of the average Danish diet (15 E% from protein, max 35 E% from fat, and max 15 E% from saturated fat).
  Interventions: Other: Dietary intervention: CHEESE (High cheese intake)
- MEAT diet (Experimental): The MEAT diet will be a diet without dairy products. In this diet cheese is mainly replaced by high-fat mixed meat products to achieve saturated fat content and protein quality similar to that of the CHEESE diet. The MEAT diet will have the same macronutrient composition as that of the average Danish diet (15 E% from protein, max 35 E% from fat, and max 15 E% from saturated fat).
  Interventions: Other: Dietary intervention: MEAT (High Meat intake)

INTERVENTIONS:
Other: Dietary intervention: CHEESE (High cheese intake)
  Arms: CHEESE diet
Other: Dietary intervention: MEAT (High Meat intake)
  Arms: MEAT diet
Other: Dietary intervention: CARB (High Carbohydrate intake)
  Arms: CARB diet

SUMMARY:
The main objective of the current study is to examine whether a high intake of regular-fat cheeses (Danbo and Cheddar) affect blood lipids differently than an isocaloric intake of either other fatty animal food products or of starchy carbohydrates. Furthermore, effects on fat digestibility, blood pressure, anthropometry, bile acid metabolism and insulin sensitivity is investigated.

To do this, a randomized crossover intervention study with 3x14 days full diet periods (cheese diet, meat diet or carb diet)will be conducted in 16 postmenopausal women. Between the diet periods there will be at least 14 days of wash-out where the subjects eat their habitual diets. Fasting blood samples will be drawn before and after the diet periods, and also a non-fasting blood sample will be drawn after the diet periods. Furthermore, total feces is collected the last 5 days of each diet period.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Postmenopausal for >1 year
* Age 45-68 years
* BMI 25-32 kg/m2
* TC > 4.5 mmol/L and < 7 mmol/L
* Systolic blood pressure <160 mmHg and/or diastolic blood pressure <100 mmHg

Exclusion Criteria:

* Chronic diseases (known diabetes; CVD; other chronic diseases which could affect the results of the present study)
* Milk allergy
* Nut allergy
* Use of dietary supplements incl. multivitamins (2 months before and during the entire study period)
* Smoking
* Elite athletes (>10 hours of strenuous physical activity per week)
* Use of prescription medicine which could affect the results of the present study including systemic glucocorticoids
* Use of lipid-lowering agents
* Stable dose of antihypertensive medication >3 months before study commencement for subjects with high blood pressure
* Hormone replacement therapy
* Blood donation <1 month before study commencement and during study period
* Simultaneous participation in other clinical studies
* Inability (physically or psychologically) to comply with the procedures required by the protocol

Ages: 45 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | day 1 and day 14 in each diet period
  fasting, mmol/l

SECONDARY OUTCOMES:
Blood lipid concentrations | day 1 and day 14 in each diet period
  Total cholesterol and HDL cholesterol. Fasting, mmol/l.
  Triglycerides. Fasting and non-fasting, mmol/l
ApoA1 and ApoB | day 1 and day 14 in each diet period
Dietary fat digestibility | During day 10-14 in each period
  Fecal fat and energy excretion.
  Total excretion of fecal fat (grams/day) and energy (kJ/day) averaged over five days
Blood pressure | day 1 and day 14 in each diet period
  mmHg
Anthropometry | day 1 and day 14 in each diet period
  waist to hip ratio, waist circumference and body weight
Insulin sensitivity | day 1 and 14 in each diet period
  Fasting and non-fasting glucose and insulin
Bile acid metabolism | day 14 of each intervention period
  Serum alpha-HC, fecal bile acid excretion

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof, MD, Principal Investigator — Head of Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Thorning TK, Raziani F, Bendsen NT, Astrup A, Tholstrup T, Raben A. Diets with high-fat cheese, high-fat meat, or carbohydrate on cardiovascular risk markers in overweight postmenopausal women: a randomized crossover trial. Am J Clin Nutr. 2015 Sep;102(3):573-81. doi: 10.3945/ajcn.115.109116. Epub 2015 Jul 15. PMID 26178720